CLINICAL TRIAL: NCT01010724
Title: A Randomized, Double-Blind, Placebo Controlled Study of Biap, an Endotoxin Detoxificating Moiety, in Patients Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass
Brief Title: Efficacy and Safety Study on bIAP
Acronym: APPIRED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Alloksys Life Sciences B.V. (Industry)
Responsible Party: Dr. J.P.A.M. Schonberger, Catharina hospital, department of Cardiothoracic surgery
Other Study IDs: APPIRED ALS-001-2005
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease; Endotoxin-mediated Complications From Cardiopulmonary Bypass Surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2-(3',4'-dihydroxyphenyl-1-azo)benzimidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bIAP (Experimental): Dosage 200 IU bIAP/kg: 1000 IU prior to anaesthesia administered as a bolus followed by intravenous continuous infusion of 5,6 IU/kg/hr for approximately 36 hours.
  Interventions: Drug: bIAP
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bIAP
  Arms: bIAP
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study drug bIAP, or matching placebo, will be administered as a bolus of 1000 Units bIAP or matching placebo prior to anaesthesia (T = -15 minutes), directly followed by intravenous continuous infusion of about 5.6 units per kg bodyweight/hr at pump rate 4 ml/hr for approximately 36 hrs (total 200 IU/kg/36 hrs) into each of a total of 50 patients scheduled for coronary artery bypass graft surgery (CABG). Risk of surgical complications and mortality due to co-morbid conditions will be collected and the EuroSCORE will be used to screen patients prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients of any race in the ages of >18 years. Women must be of non-childbearing potential.
2. Patients scheduled for coronary artery bypass surgery with CPB.
3. Patients must have a EuroSCORE (Appendix I) of >2 and <6.
4. Patients who have given written informed consent prior to participation in the trial and who undertake to comply with the protocol.

Exclusion Criteria:

1. Patients who are unwilling or unable to be fully evaluated for follow-up.
2. Patients who undergo CABG for emergency due to complications from percutaneous transluminal coronary angioplasty (PTCA)/ catheterization, unstable angina or ongoing myocardial infarction.
3. Patients who have base alkaline phosphatase levels at > 100 IU/l (70 IU/L as mean concentration) levels, or levels < 30 IUnits/L (ammediol, DEA units)

   (values base levels in glycine units at pH9.6 and 25 C are respectively >40 and < 12 IU/L).
4. Patients who show pre-operative infections or who are suspected of having endocarditis or systemic infection.
5. Patients who refuse to accept medically-indicated blood products.
6. Patients who have evidence of significant hepatic disease, including history of clinical signs or laboratory values of total bilirubin > 2.0 mg/dL, ALT or AST> 3X upper limit of normal.
7. Patients who received investigational drugs in the 30 days prior to study drug administration, or are currently participating in a study during which the administration of investigational drugs within one month is anticipated.
8. Patients who require pre-operative ventilatory support.
9. Patients who have renal insufficiency (history of creatinine> 2.0 mg/dL) or chronic renal failure requiring dialysis.
10. Patients who are planned to receive leukocyte-depletion filtration as part of the bypass circuitry.
11. Patients with severe neurological deficits (see Appendix I).
12. Patients who have a recent history of substance or alcohol abuse.
13. Patients with a diagnosis of idiopathic thrombocytopenia.
14. Concomitant surgical procedures (i.e., not included in Appendix VI) anticipated to require greater than 2.5 hours time "on-pump" or patients for whom surgery other than coronary artery bypass surgery is planned during the 30-day study period.
15. Patients with a history of cancer who have received chemotherapy or radiation therapy within the past 3 months. Patients receiving only adjuvant hormonal therapy are not excluded. If the cancer has not resolved completely, the patient should not be enrolled without permission of Alloksys.
16. Patients who are scheduled to receive "stress doses" of glucocorticoids (i.e., doses >2 mg/kg/day of methylprednisolone or equivalent) prior to, during or following the operation.
17. Patients who are vegetarians or vegenists or those patients that may be expected not to be tolerant for bovine proteins.
18. Patients who have a BMI (body mass index) < 18 or > 30
19. Patients who are, in the opinion of the Investigator or the Sponsor, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To determine the efficacy and safety of bIAP as a prophylaxis against endotoxin-mediated complications from cardiopulmonary bypass surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina hospital, dept. of Cardiothoracic Surgery, Eindhoven, Netherlands